CLINICAL TRIAL: NCT01118117
Title: A Multi-center Clinical Trial of the Misago™ Self-Expanding Stent System for Superficial Femoral Artery
Acronym: OSPREY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Medical Corporation (Industry)
Collaborators: ClinLogix. LLC (Industry); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIS2009-02
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Vascular Disease
Keywords: atherosclerotic stenosis; occlusions; Superficial Femoral Artery; SFA
MeSH Terms: conditions — Peripheral Vascular Diseases; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Misago™ Self-Expanding Stent System (Experimental)
  Interventions: Device: Misago™ Self-Expanding Stent System

INTERVENTIONS:
Device: Misago™ Self-Expanding Stent System — Transcatheter placement of an intravascular stent(s)
  Other Names: Misago; OSPREY

SUMMARY:
OSPREY is a multi-center, single arm, non-randomized, prospective clinical trial. Subjects will undergo a superficial femoral artery (SFA) stent procedure using the Misago™ Peripheral Self Expanding stent once all of the inclusion and none of the exclusion criteria are met. The stent efficacy and safety will be evaluated immediately post procedure, and at 30 days, 6, 12, 24, and 36 months post procedure. A subject is considered enrolled into the OSPREY study after he/she signs the informed consent and meets all inclusion/exclusion criteria.

The study objectives are to demonstrate that efficacy and safety of this novel stent design are not inferior to historical Percutaneous Transluminal Angioplasty (PTA) and stent outcomes and meet the performance goals as published in the objective performance goals by Rocha-Singh, et al. This is a multi-center, single arm, non-randomized, prospective clinical trial of the Misago™ Self-Expanding Stent System for the treatment of atherosclerotic stenosis and occlusions of the SFA. The primary endpoint of stent patency will be evaluated at 12 months.

ELIGIBILITY:
Inclusion Criteria:

Pre-procedure:

1. Female or male age greater than or equal to 18 years and of legal consent.
2. Subjects must be willing to comply with the specified follow-up evaluation schedule.
3. Informed consent (signed and dated) prior to any study-related evaluation or procedures.
4. Symptomatic leg ischemia without tissue loss by Rutherford classification (category 2, 3 or 4).
5. Resting ABI of <0.9, or abnormal exercise ABI.
6. De novo lesion(s) (one or multiple lesions) with >50% stenosis, or occlusion which require treatment, and a total lesion length of >40 mm and <150 mm of the above-the-knee SFA in one limb. The target lesion should be treatable with no more than two overlapping stents, minimizing the stent overlap up to 10 mm (by visual estimate).
7. All lesions are at least 3 cm above the knee joint, defined as the distal end of the femur at the knee joint, and at least 2 cm distal to the origin of the profunda artery.
8. Reference vessel diameter of >4.0 mm and <7.0 mm.
9. Target lesion length of > 40 mm and <150 mm.
10. Patent popliteal artery (no stenosis > 50%) and at least one patent tibioperoneal run-off vessel with < 50% stenosis confirmed by angiography within 30 days of enrollment.

Exclusion Criteria:

1. Pre-existing autoimmune disease.
2. Pre-existing terminal illness with life expectancy of less than three (3) years.
3. Participation in another investigational device or therapeutic intervention trial within the past three (3) months.
4. Previous enrollment in this study.
5. Previous bypass surgery or stenting in the SFA or distally.
6. Scheduled for a staged procedure to treat lesions within the aorta or run-off after enrollment.
7. Co-existing aneurysmal disease of the aorta, iliac artery, SFA, or popliteal arteries requiring treatment.
8. Any inflow disease of the ipsilateral pelvic arteries (more than 50 percent stenosis or occlusion) that has not been treated prior to enrollment (Treatment of iliac arteries before SFA intervention is permitted, except for common femoral stenosis).
9. A recent (< 6 week) history of clinically significant gastrointestinal bleeding, major surgery, myocardial infarction or untreated coagulopathy.
10. Known sensitivity or allergy to aspirin, radiographic contrast agents (that cannot be pre-treated adequately), nitinol, gold, or both heparin and bivalirudin.
11. Angiographic evidence of acute thrombus.
12. Sudden worsening of symptoms in the last 30 days.
13. Subjects with acute/chronic renal dysfunction or estimated glomerular filtration rate (eGFR) <30 ml/min. Chronic hemodialysis subjects are not eligible for this protocol.
14. Severe calcification or excessive tortuosity at target lesion.
15. Subjects unable to tolerate anticoagulant therapy or antiplatelet therapy.
16. Women who are currently pregnant. (A negative pregnancy test for female subjects of child bearing potential is required).
17. The target lesion(s) cannot be successfully crossed with a guide wire.*
18. Lower extremity deep venous thrombosis in the study limb within the prior 30 days.
19. Chronic venous disease with active or recent (< 30 day) skin ulceration.
20. Known or suspected active systemic infection.
21. Two (2) months previous history of non-hemorrhagic stroke and or history of hemorrhagic stroke.
22. Treatment that requires access via upper extremity, popliteal artery, or pedal artery.
23. Evidence of severe or uncontrolled systemic disease of any condition which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
24. Use of re-entry, ablative, or atherectomy devices to cross the lesion.*

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Angle, MD, Principal Investigator — University of Virginia
Locations (31):
- United States (31):
  - University Of Alabama, Birmingham, Alabama
  - Cardiology Associates of Mobile, Fairhope, Alabama
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Long Beach VA Healthcare Center, Long Beach, California
  - Christiana Care, Newark, Delaware
  - Bradenton Cardiology Center, Bradenton, Florida
  - Florida Research Network, Gainesville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Coastal Vascular and Interventional, PLLC, Pensacola, Florida
  - Cardiovascular Associates, Elk Grove Village, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa Healthcare, Iowa City, Iowa
  - Kings Daughters Medical Center, Ashland, Kentucky
  - Michigan Heart, Ypsilanti, Michigan
  - Hunterdon Cardiovascular Associates, Flemington, New Jersey
  - Columbia University Medical Center, New York, New York
  - Hillsboro Cardiology, Hillsboro, Oregon
  - Central Bucks Specialists, Doylestown, Pennsylvania
  - St. Mary Medical Centere Research Institute, Langhorne, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Berks Cardiologists, Ltd, Wyomissing, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Premier Clinical Reesearch, Knoxville, Tennessee
  - East Tennessee Cardiovascular Research-Turkey Creek Medical Center, Knoxville, Tennessee
  - Amarillo Heart Clinical Research Institute, Amarillo, Texas
  - University of Virginia, Charlottesville, Virginia
  - Centra Cardiovascular Group, Lynchburg, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Columbia- St. Mary's, Milwaukee, Wisconsin

REFERENCES:
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972
- [Derived] Ohki T, Angle JF, Yokoi H, Jaff MR, Popma J, Piegari G, Kanaoka Y; OSPREY investigators. One-year outcomes of the U.S. and Japanese regulatory trial of the Misago stent for treatment of superficial femoral artery disease (OSPREY study). J Vasc Surg. 2016 Feb;63(2):370-6.e1. doi: 10.1016/j.jvs.2015.08.093. Epub 2015 Oct 17. PMID 26483003
- [Derived] Schulte KL, Kralj I, Gissler HM, Bagnaschino LA, Buschmann I, Pernes JM, Haage P, Goverde P, Beregi JP, Valka M, Boudny J, Geibel T, Velkoborsky M, Zahringer M, Paetzel C, Fanelli F, Muller-Hulsbeck S, Zeller T, Langhoff R. MISAGO 2: one-year outcomes after implantation of the Misago self-expanding nitinol stent in the superficial femoral and popliteal arteries of 744 patients. J Endovasc Ther. 2012 Dec;19(6):774-84. doi: 10.1583/JEVT-12-3861MR.1. PMID 23210876

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 261 subjects were enrolled in the pivotal study cohort. An additional 15 subjects were implanted with a single, 150mm stent as part of a long length stent (LL) sub-study. The LL sub-study included safety data through 30 days post-procedure and was analyzed separately from the pivotal study cohort.
Groups:
- Misago™ Self-Expanding Stent System: Subjects received treatment with the Misago™ Self-Expanding Stent
- Long Length Stent Sub-Study Cohort: Misago™ Self-Expanding Stent System: Transcatheter placement of a single, 150 mm intravascular stent
Period: Overall Study
Arm/Group | Misago™ Self-Expanding Stent System | Long Length Stent Sub-Study Cohort
Started | 261 | 15
Completed | 240 | 15
Not Completed | 21 | 0
Not completed — Death | 8 | 0
Not completed — Lost to Follow-up | 6 | 0
Not completed — Missed 12 Month Visit | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Long Length (150mm) Misago™ Self-Expanding Stent System: Misago™ Self-Expanding Stent System: Transcatheter placement of a single, 150mm intravascular stent
- Total: Total of all reporting groups
Arm/Group | Misago™ Self-Expanding Stent System | Long Length (150mm) Misago™ Self-Expanding Stent System | Total
Number analyzed (Participants) | 261 | 15 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (10) | 70.7 (10.9) | NA (NA) — Combined analysis of pivotal cohort and LL sub-study cohort was not completed
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 8 | 100
  Male | 169 | 7 | 176
Region of Enrollment [Number; unit: participants]
  United States | 201 | 15 | 216
  Japan | 50 | 0 | 50
  Taiwan | 9 | 0 | 9
  Korea, Republic of | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: The primary effectiveness endpoint was defined as stent patency at 12 months as evidenced by absence of TLR and a peak systolic velocity ratio < 2.0 from DUS obtained within the 12 months visit window.
Time Frame: 12 Months post-procedure
Population: Analysis comprised of 261 subjects enrolled in pivotal trial and missing data imputed as loss of patency under the intention-to-treat (ITT) analysis. Study success was based on the proportion of patients with stent patency when tested against a performance goal of 66% using the lower bound of the 95% confidence interval.
Measure: Number (95% Confidence Interval); unit: percentage of stent patency
Groups:
- Non-Randomized: Misago™ Self-Expanding Stent System: Transcatheter placement of an intravascular stent(s)
Arm/Group | Non-Randomized
Number analyzed (Participants) | 261
percentage of stent patency | 54.0 [48.0 to 60.0]

2. Secondary Outcome: Primary Effectiveness Endpoint in Modified Intent-to-Treat (mITT) Cohort
Description: Primary effectiveness endpoint was defined as absence of TLR and stent patency at 12 months as evidenced by a peak systolic velocity ratio < 2.0 from DUS obtained within the 12 months visit window. Because patency beyond the 12 months visit window may be considered as patency at 12 months, the out-of-window patency is imputed as treatment success. The modified intention to treat (mITT) cohort had 226 subjects (excluded subjects with unknown primary effectiveness endpoint).
Time Frame: 12 Months post-procedure
Population: The modified intention to treat (mITT) cohort had 226 subjects (excluded subjects with unknown primary effectiveness endpoint).
Measure: Number; unit: percentage of stent patency
Arm/Group | Non-Randomized
Number analyzed (Participants) | 226
percentage of stent patency | 62.4

3. Primary Outcome: Primary Safety Endpoint
Description: The primary safety endpoint for this study was freedom from major adverse events (MAE) at 30 days post-procedure. MAE was defined as TLR, amputation of the treated limb, or death.
Time Frame: 30 days post-procedure
Population: Study success was based on the proportion of patients with freedom from MAE at 30 days post-procedure when tested against a performance goal of 88% using the lower bound of the 95% confidence interval. In both cohorts, the lower confidence interval exceeded the prespecified performance goal indicating the study met its primary safety endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects without a MAE
Groups:
- Long Length Stent Sub-Study Cohort: Misago™ Self-Expanding Stent System: Transcatheter placement of a single, 150mm intravascular stent
Arm/Group | Non-Randomized | Long Length Stent Sub-Study Cohort
Number analyzed (Participants) | 261 | 15
percentage of subjects without a MAE | 99.2 [97.1 to 100] | 100 [92.8 to 100]

4. Secondary Outcome: Primary Effectiveness Endpoint Using a Peak Systolic Velocity Ratio of ≤ 2.4 (i.e., Modified VIVA Criteria) in the mITT Cohort
Description: The primary effectiveness endpoint was defined as absence of TLR and stent patency at 12 months as evidenced by a peak systolic velocity ratio < 2.0 from duplex ultrasound. Additional considerations were made using a more contemporary approach to evaluate stent patency using a peak systolic velocity ratio (PSVR) ≤ 2.4 (i.e., modified VIVA criteria). This outcome evaluated the modified intent-to-treat (mITT) cohort comprised of 226 subjects (excluded subjects with unknown primary effectiveness endpoint)
Time Frame: 12 Months post-procedure
Population: Analysis uses a more contemporary approach to evaluate primary stent patency using a peak systolic velocity ratio ≤ 2.4 (modified VIVA criteria). Because patency beyond the 12 months visit window may be considered as patency at 12 months, the out-of-window patency is imputed as treatment success in the analysis.
Measure: Number; unit: percentage of stent patency
Arm/Group | Non-Randomized
Number analyzed (Participants) | 226
percentage of stent patency | 69.9

5. Secondary Outcome: Occurrence of Target Lesion Revascularization
Description: The occurrence of clinically driven Target Lesion Revascularization (TLR) was measured at 12 months post-procedure.
  Clinically driven defined as:
  * More than 50 percent stenosis with worsening symptoms, OR
  * More than 70 percent stenosis without symptoms
Time Frame: 12 Months post-procedure
Population: Comprised of all subjects enrolled in the pivotal OSPREY trial (N=261)
Measure: Number; unit: percentage of subjects with TLR
Arm/Group | Non-Randomized
Number analyzed (Participants) | 261
percentage of subjects with TLR | 13.0

6. Secondary Outcome: Device Related Peri-Procedural Complications
Description: Peri-procedural (prior to discharge) measure of success (i.e., patency and none of the following: death, stroke, MI, embolization, thrombosis, and occlusion)
Time Frame: Prior to Hosptial Discharge
Population: All enrolled participants evaluated prior to hospital discharge
Measure: Number; unit: percentage of subjects with event
Arm/Group | Non-Randomized
Number analyzed (Participants) | 261
percentage of subjects with event | 2.3

7. Secondary Outcome: Technical Success
Description: Technical Success defined by the following conditions:
  * Successful delivery of the stent at the lesion site
  * Stent(s) successfully deployed in lesion with adequate lesion coverage
Time Frame: Intra-procedure
Population: All subjects enrolled in pivotal trial
Measure: Number; unit: percentage of subjects with success
Arm/Group | Non-Randomized | Long Length Stent Sub-Study Cohort
Number analyzed (Participants) | 261 | 15
percentage of subjects with success | 100 | 93.3

8. Secondary Outcome: Procedural Success
Description: Procedural success defined as: attainment of < 30% residual stenosis of the target lesion and no peri-procedural complications defined as: death, stroke, myocardial infarction, emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel
Time Frame: Intra-procedure
Measure: Number; unit: percentage of subjects with success
Arm/Group | Non-Randomized | Long Length Stent Sub-Study Cohort
Number analyzed (Participants) | 261 | 15
percentage of subjects with success | 93.5 | 100

9. Secondary Outcome: Clinical Success
Description: Clinical success defined as: relief or improvement from baseline symptoms as measured by the Rutherford score for chronic limb ischemia at 30 days as compared to baseline
Time Frame: 30 days post-procedure
Measure: Number; unit: percentage of subjects with success
Arm/Group | Non-Randomized | Long Length Stent Sub-Study Cohort
Number analyzed (Participants) | 260 | 14
percentage of subjects with success | 90.0 | 92.9

10. Secondary Outcome: Major Adverse Events (MAEs) Through 12 Months Post-procedure
Description: The incidence of MAEs occurring within 12 months of the procedure. MAE is defined as target lesion revascularization (TLR), amputation of the treated limb, or death.
Time Frame: 12 Months post-procedure
Measure: Number; unit: percentage of subjects with event
Arm/Group | Non-Randomized
Number analyzed (Participants) | 261
percentage of subjects with event | 16.1

11. Secondary Outcome: Stent Fracture at 12 Months
Description: Occurrence of stent fracture as determined by core laboratory analysis
Time Frame: 12 Months post-procedure
Population: X-rays for 324 stents (234 subjects) were available for analysis by the angiographic core laboratory to evaluate stent fractures at 12 months post-procedure. One stent fracture was caused by a physician during a non-study peripheral intervention.
Measure: Number; unit: percentage of fracture occurrence
Units Other Than Participants: stents
Arm/Group | Non-Randomized
Number analyzed (Participants) | 234
Number analyzed (stents) | 324
percentage of fracture occurrence | 0.9

ADVERSE EVENTS:
Time Frame: For the pivotal study cohort, adverse events from enrollment through study completion (12 months post-procedure) are presented. For the long length stent sub-study, adverse events from enrollment through 30 days are presented.
Arm/Group | Non-Randomized | Long Length Stent Sub-study Cohort
Serious Adverse Events (participants affected / at risk) | 135/261 | 1/15
Other Adverse Events (participants affected / at risk) | 167/261 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Randomized (N=261) | Long Length Stent Sub-study Cohort (N=15)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 6 | 0
Angina Pectoris (Cardiac disorders) | 4 | 0
Angina Unstable (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 5 | 0
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 7 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Pericarditis Constrictive (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Amaurosis Fugax (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Impaired Gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Mesenteric Artery S'tenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Device Failure (General disorders) | 1 | 0
Device Occllusion (General disorders) | 3 | 0
Generalised Oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 0
Cholecystitis Infective (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Graft Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 0
Post-Operative Wound Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 1 | 0
Arterial Restenosis (Injury, poisoning and procedural complications) | 4 | 0
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 30 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Pulse Absent (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance Disorder (Nervous system disorders) | 1 | 0
Brain stem Stroke (Nervous system disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 3 | 0
Carotic Artery Disease (Nervous system disorders) | 2 | 0
Cerbral haemorrhage (Nervous system disorders) | 1 | 0
Cerbral Infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 3 | 0
Essential Tremor (Nervous system disorders) | 1 | 0
Lacunar Infarction (Nervous system disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 7 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial Thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Extremity Necrosis (Vascular disorders) | 1 | 0
Femoral Artery Dissection (Vascular disorders) | 1 | 0
Femoral Artery Occlusion (Vascular disorders) | 4 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypertensive Emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 0
Iliac Artery Occlusion (Vascular disorders) | 2 | 0
Intermittent Claudication (Vascular disorders) | 15 | 0
Ischaemic Limb Pain (Vascular disorders) | 1 | 0
Peripheral Artercy Occlusive Disease (Vascular disorders) | 2 | 0
Peripheral Artery Stenosis (Vascular disorders) | 11 | 0
Peripheral Embolism (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 5 | 0
Subclavian Artery stenosis (Vascular disorders) | 1 | 0
Vascular Pseudoaneurysm (Vascular disorders) | 1 | 0
Right Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Randomized (N=261) | Long Length Stent Sub-study Cohort (N=15)
Anaemia (Blood and lymphatic system disorders) | 13 | 0
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 41 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 21 | 0
Pain in Exteremity (Musculoskeletal and connective tissue disorders) | 14 | 0
Haematoma (Vascular disorders) | 13 | 0
Hypertension (Vascular disorders) | 22 | 0
Intermittent Claudication (Vascular disorders) | 27 | 0
Peripheral Artery Stenosis (Vascular disorders) | 16 | 0
Post Dilatation Dissection (Vascular disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Allergy to Vancomycin (Immune system disorders) | 0 | 1
Rash-waist to knees (Skin and subcutaneous tissue disorders) | 0 | 1
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1
Burning Right Leg (Nervous system disorders) | 0 | 1
bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
hypertension post-procedure (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less